CLINICAL TRIAL: NCT05534152
Title: The Effect of Consumption of Sumac in Vegetable Soup on Appetite and Food Intake Among Older Adults (Aged Over 65 Years) and Young Adults (Aged 18-35 Years)
Brief Title: Effect of Sumac on Appetite and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UREC 181174
Record Dates: First submitted 2022-07-31; First posted 2022-09-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Appetite; Food Intake

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soup with no sumac (Placebo Comparator): 150 g butternut squash soup with no added sumac
  Interventions: Other: sumac
- Sumac added to soup at the end of cooking (Experimental): 150 g butternut squash soup with 1% sumac added at the end of cooking
  Interventions: Other: sumac
- Sumac added to the sumac during cooking (Experimental): 150 g butternut squash soup with 1% sumac added during cooking
  Interventions: Other: sumac

INTERVENTIONS:
Other: sumac — 1% iranian brown sumac

SUMMARY:
Sumac, is a spice that is widely used in Turkish, Iranian and Middle Eastern foods. In these regions, the fruit of sumac is used for seasoning or flavouring, as an appetizer and for souring food. This spice has also been used in herbal folk medicine to relieve certain conditions including bowel disorders, anorexia and indigestion. In addition, many studies have shown that sumac contains a high level of antioxidant activity and polyphenol content that may benefit certain diseases such as cancer and diabetes. The aim of this study was to assess the level of the appetite and food intake among young adults in comparison with free living older adults following the consumption of sumac. This was achieved by assessing the amount of food intake during a lunch course and the impact on food intake for the subsequent 12 hours.

DETAILED DESCRIPTION:
Rhus coriaria Linn, also known as Sumac, is a spice that is widely used in Turkish, Iranian and Middle Eastern foods. In these regions, the fruit of sumac is used for seasoning or flavouring, as an appetizer and for souring food. This spice has also been used in herbal folk medicine to relieve certain conditions including bowel disorders, anorexia and indigestion. In addition, many studies have shown that sumac contains a high level of antioxidant activity and polyphenol content that may benefit certain diseases such as cancer and diabetes.

Taste and smell perception may play a vital role in food preference, nutrient intake and appetite; however, both ageing and disease can have a negative impact on these senses. It has been suggested that by 2025 the older adult population (i.e. those aged 60years and over) worldwide will rapidly increase and reach 1.12 billion. One of the major physiological changes in this age group is the loss or reduction in sensory perception including smell and taste. These changes as a result of ageing and medication increase the risk of poor health by reducing the enjoyment of food followed by decreasing food and nutrient intake.

It is possible, therefore, that all these factors together may lessen the enjoyment of food, leading to malnutrition and disease complications. In light of the above, the aim of this study was to assess the level of the appetite and food intake among young adults in comparison with free living older adults following the consumption of sumac. This was achieved by assessing the amount of food intake during a lunch course and the impact on food intake for the subsequent 12 hours.

This study assessed the use of sumac at 1% dose (0.37g) of total volume of a vegetable soup (150g), in two forms: 1) added to finished cooked soup 2) added to the soup from the beginning of the cooking process, in addition to consumption of the same soup without added sumac as the control soup. The study comprised of 20 young adults (18-35 years old) and 20 free living older adults aged >65 years. Each participant in these groups attended the Oxford Brookes Centre for Nutrition and Health (OxBCNH) for three sessions and each session lasted up to one hour.

ELIGIBILITY:
Inclusion Criteria:

* • Adults, aged >65 years

  * Adults, 18-35 years
  * No allergy to any herbs and spices
  * No allergy to vegetables including celery and tomato
  * Non-smoker
  * Do not have a cold or hay fever (on test day)
  * No medication that may affect the sensory taste such as: antibiotics, antihistamines and decongestants, anti-inflammatory agents, and muscle relaxants (Bromley, 2000)
  * Ability to read and understand written information in English
  * Ability to attend, stand and sit for up to one hour
  * The normal level of capability of functional activity (i.e. traveling out to the neighbourhood, shopping alone)
  * Not diagnosed with Dementia

Exclusion Criteria:

* Disease that may affect the taste and smell sensation including local chronic or acute inflammatory nasal disease and oral and perioral infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Energy intake in kilojoules and kilocalories | 9 hours
  Energy intake at an ad libitum lunch after the soup and for the rest of the day using Nutritics dietary assessment software.
Carbohydrate intake in grams | 9 hours
  Carbohydrate intake at an ad libitum lunch after the soup and for the rest of the day using Nutritics dietary assessment software.
Protein intake in grams | 9 hours
  Protein intake at an ad libitum lunch after the soup and for the rest of the day using Nutritics dietary assessment software.
Fat intake in grams | 9 hours
  Fat intake at an ad libitum lunch after the soup and for the rest of the day using Nutritics dietary assessment software.
Amount of food consumed at lunch in grams | 9 hours
  Amount of food (pasta) consumed in grams at the ad libitum lunch

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No